CLINICAL TRIAL: NCT07136896
Title: Nutritional Assessment of Patient of Mucopolysaccharide
Brief Title: Nutritional Assessment in Patient of Mucopolysaccharide "
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Sayed Abdelbaseer, Principal Investigator,, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mucopolysacharidosis
Record Dates: First submitted 2025-08-09; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Mucopolysaccharidosis (MPS); Malnutrition (Calorie); Undernutrition
Keywords: Caloric deficiency; Pediatric nutrition
MeSH Terms: conditions — Mucopolysaccharidoses; Malnutrition

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel groups: children with mucopolysaccharidosis (MPS) and age-matched healthy controls. Both groups will undergo the same nutritional assessment protocol for comparison.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Assessment in Children with Mucopolysaccharidosis (Other): Participants diagnosed with Mucopolysaccharidosis will undergo detailed nutritional assessment, including anthropometric measurements, skinfold thickness evaluation, and bioelectrical impedance analysis. Dietary intake will be recorded, and relevant biochemical parameters will be measured.
  Interventions: Other: Nutritional Assessment Protocol

INTERVENTIONS:
Other: Nutritional Assessment Protocol — Participants will undergo a comprehensive nutritional assessment, including anthropometric measurements (weight, height, BMI, skinfold thickness), dietary intake evaluation through 24-hour recall, and bioelectrical impedance analysis to assess body composition. Relevant biochemical parameters will also be measured to evaluate nutritional status

SUMMARY:
" Nutritional assessment in patients of Mucopolysaccharide "

DETAILED DESCRIPTION:
The mucopolysaccharidoses (MPS) are lysosomal diseases caused by the deficiency of enzymes required for the stepwise breakdown of glycosaminoglycans (GAGs), previously known as mucopolysaccharides, Fragments of partially degraded GAGs accumulate in the lysosomes, resulting in cellular dysfunction and clinical abnormalities The main GAG chains are degraded by 11 lysosomal hydrolases enzymes gives rise to the progressive accumulation of GAGs in most tissues and organ systems, as well as in urine Individuals with MPS disorders share many similar symptoms such as multiple organ involvement, distinctive "coarse" facial features, and abnormalities of the skeleton especially joint problems. Additional findings include short stature, heart abnormalities, breathing irregularities, hepatosplenomegaly and neurological abnormalities. The severity of the different MPS disorders varies greatly among affected individuals, even among those with the same type of MPS and even among individuals of the same family.

In most cases of MPS, affected infants appear normal at birth and symptoms become apparent around the age of one or two, however, in MPS VII, approximately 40% of pregnancies with an affected baby are complicated by a condition called non-immune hydrops fetalis. Mild forms of these disorders may not become apparent until childhood or adolescence. In most cases, the mucopolysaccharidoses are chronic, progressive disorders and, depending upon the type of MPS and severity, affected individuals may experience a decline in physical and mental function, sometimes resulting in life-threatening complications.

Nutritional assessment in MPS focuses on identifying and addressing potential deficiencies and challenges related to the disease's impact on growth, development, and feeding. This involves evaluating dietary intake, assessing growth parameters, and monitoring for specific nutrient deficiencies, particularly those impacting bone health and overall metabolic function The dietetic treatment of MPS does not only aim to correct diarrhea and constipation but also help in the consistency of the dysphagia treatment probable adequacy in vitamin (B1, B2, and B3) levels since they are largely spread in the food. These vitamins may participate in energetic metabolism, in redox reactions. In this regard, niacin plays a critical role in nucleic acids, fatty acids and cholesterol synthesis, DNA repair, and steroid hormones production.

ELIGIBILITY:
Inclusion Criteria:Confirmed diagnosis of mucopolysaccharidosis (any subtype) by enzymatic assay or genetic testing

Age between 1 and 18 years

Stable clinical condition at time of enrollment

Informed consent obtained from parent/guardian, and assent from child when applicable -

Exclusion Criteria:Presence of other chronic conditions affecting growth or nutrition (e.g., untreated endocrine disorders, severe cardiac failure unrelated to MPS)

Acute illness or hospitalization within the last 2 weeks prior to assessment

Patients who received nutritional supplementation or dietary intervention within 3 months prior to enrollment that could affect baseline nutritional assessment

Refusal or inability to comply with study assessments

-

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-16 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of malnutrition among patients with mucopolysaccharidosis | 1 year
  The percentage of patients diagnosed with malnutrition, as determined using the World Health Organization (WHO) growth standards. Malnutrition will be defined based on weight-for-age, height-for-age, and weight-for-height Z-scores below -2 standard deviations. Data will be collected at baseline and expressed as a percentage of the study population.
severity of malnutrition among patients with mucopolysaccharidosisby WHO growth standards Z-scores (weight-for-age, height-for-age, weight-for-height) | At baseline (upon enrollment)
  Severity of malnutrition will be assessed using the Gomez classification based on weight-for-age percentage of the median for the reference population. Categories include: mild (75-89%), moderate (60-74%), and severe (<60%). Data will be expressed as the proportion of patients in each severity category at baseline
Prevalence and severity of malnutrition among patients with mucopolysaccharidosis | At baseline (upon enrollment)
  The proportion of patients diagnosed with mucopolysaccharidosis (MPS) who present with any degree of malnutrition, categorized as mild, moderate, or severe according to WHO growth standards. Severity will be determined using anthropometric indices (weight-for-age, height-for-age, BMI-for-age z-scores, and mid-upper arm circumference) and compared across disease subtypes and age groups.